CLINICAL TRIAL: NCT02252952
Title: A Comparison of the Effects of Sugar Sweetened Beverages (SSBs), Diet Beverages and Water on Weight, Body Composition, Liver and Muscle Fat Infiltration, Visceral Fat, Neurocognitive Function, Blood Lipids, Insulin Resistance and Hydration Status in Healthy Weight and Overweight, Premenopausal Females Aged 20-50
Brief Title: The Effect of Sugar Sweetened and Diet Beverages Consumed as Part of a Weight-Maintenance Diet on Fat Storage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rippe Lifestyle Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1136635
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Focus: Understanding the Obesogenic Potential of Sugars and Non-caloric Sweeteners
Keywords: Sugar Sweetened Beverages, Diet Beverages, ectopic fat, Functional MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sugar Sweetened Beverages (Experimental): Any beverage from a range of caffeine free, sugar sweetened drinks. One serving =12oz. Two servings will be consumed daily as part of a structured, weight maintenance diet for 6 months.
  Interventions: Other: Beverage Consumption
- Diet Beverage (Experimental): Any beverage from a range of caffeine free drinks sweetened with non-caloric sweetener. One serving =12oz. Two servings will be consumed daily as part of a structured, weight maintenance diet for 6 months.
  Interventions: Other: Beverage Consumption
- Water (Active Comparator): 12 oz of water. Two servings will be consumed daily as part of a structured, weight maintenance diet for 6 months.
  Interventions: Other: Beverage Consumption

INTERVENTIONS:
Other: Beverage Consumption

SUMMARY:
The purpose of this study is to investigate the effects of consumption of sugar sweetened and diet beverages on overall fat mass and the fat mass of various tissues implicated in the dysregulation of glucose metabolism. In addition, hypothalamic activity will also be investigated after acute exposure to sugar sweetened and diet beverages, and again after 6 months of daily consumption.

DETAILED DESCRIPTION:
Excess fat deposition in skeletal muscle and the liver have both been implicated in the metabolic dysregulation that leads to type II diabetes. It has been shown that daily consumption of sugar sweetened beverages can lead to increases in the fat mass of these organs. However, little appreciation was given for the effect of overall changes in weight and fat mass or how applicable the doses provided may be for how sugar sweetened beverages are typically consumed.

In addition, it has recently been shown that sugars can suppress hypothalamic activity and alter patterns of brain connectivity in regions known to be involved in homeostasis and reward aspects of food intake. However, these observations were made after large doses or sugars not commonly consumed in isolation from other sugars or other macronutrients. Foods containing non-caloric sweeteners have also been suggested to suppress hypothalamic activity due to the disconnect between perceived sweetness and calories consumed.

AIM 1: To investigate the response to six months of daily consumption of sugar sweetened or diet beverages as part of a weight-stable structured diet on whole body fat content, but also specifically fat content of the liver, skeletal muscles the abdomen.

AIM 2: To investigate hypothalamic activity after acute exposure to sugar sweetened and or diet beverages, and whether chronic exposure for 6 months induces any changes in hypothalamic activity.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age between 20-50 years
* Body Mass Index (BMI) 21.0 to less than 30.0
* Consumer of at least one sugar sweetened or diet beverage per day

Exclusion Criteria:

* More than a 3% change in weight within the 3 months prior to enrollment in the study.
* Menstrual cycle that is not regular or post-menopausal
* Continued consumption of a prescription medication for weight loss. If subject is willing to discontinue prescription medication(s) immediately and willing to refrain from taking medication(s) for duration of study, he/she may be enrolled after a four-week washout period.
* Continued consumption of over-the-counter weight loss supplement(s). If subject is willing to discontinue supplement(s) immediately and willing to refrain from taking supplement(s) for duration of study, he/she may be enrolled after a two-week washout period.
* Continued enrollment in commercial weight loss program (e.g. Jenny Craig, Weight Watchers) or self-help group (e.g. TOPS, Overeaters Anonymous). If subject is willing to discontinue program immediately and willing to refrain from program for duration of study, he/she may be included after a two-week washout period.
* History of thyroid disease, but not taking medication or medication dosage changed one or more times over last 6 months. History of thyroid disease and on a stable dose of prescription medication for 6 months or longer is acceptable.
* Diagnosed with Type I or Type II diabetes or prediabetes.
* History of major surgery within three months of enrollment.
* History of heart problems (e.g. angina, bypass surgery, MI, etc.) within three months prior to enrollment.
* Presence of implanted cardiac defibrillator or pacemaker.
* Hypertension/high blood pressure, or any hypertensive medication.
* History of a surgical procedure for weight loss at any time (e.g. gastroplasty, gastric by-pass, gastrectomy or partial gastrectomy).
* Gastrointestinal disorders including chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, chronic diarrhea or active gallbladder disease.
* History of inflammatory bowel disease
* History of fatty liver
* History or presence of cancer. Persons with successfully resected basal cell carcinoma of the skin may be enrolled if treatment completed more than 6 months prior to enrollment.
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia nervosa or binge eating disorder.
* Women who are pregnant, lactating or trying to become pregnant.
* Any change in prescription medication within 3 months prior to enrollment
* Currently consuming >14 alcoholic drinks (1 drink = 12 fl oz beer, 4 fl oz wine or 1.5 fl oz liquor) per week.
* Known allergy to high fructose corn syrup, sucrose, fructose or glucose.
* History of alcohol dependency
* Extreme exercise regimes (eg. Marathon or triathlon)
* Currently smoking cigarettes
* Any clinically significant food allergy
* Participation in another clinical trial within 30 days prior to enrollment.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Fat Storage | Baseline and 6 Months
  Changes in total body adiposity (body fat percentage and fat mass) as measured by Dual X Ray Absorbance after 6 months of daily consumption of sugar sweetened or diet beverages as part of a weight-maintenance structured diet. Changes in fat content of skeletal muscle (via MRI) and liver and the abdomen (both MRS) will also be assessed.

SECONDARY OUTCOMES:
Hypothalamic Activity | 6 Months
  Hypothalamic activity in response to consumption of sugar sweetened or diet beverages consumed as part of a standardized, mixed nutrient meal will be measured by functional MRI. Changes from baseline (mean percent signal change) will be determined after 6 months of daily consumption of the test beverage

CONTACTS AND LOCATIONS:
Overall Officials: James M Rippe, MD, Principal Investigator — Rippe Lifestyle Institute
Locations (1):
- Rippe Lifestyle Institute, Celebration, Florida, United States

REFERENCES:
- [Derived] Lohner S, Kuellenberg de Gaudry D, Toews I, Ferenci T, Meerpohl JJ. Non-nutritive sweeteners for diabetes mellitus. Cochrane Database Syst Rev. 2020 May 25;5(5):CD012885. doi: 10.1002/14651858.CD012885.pub2. PMID 32449201